CLINICAL TRIAL: NCT05374642
Title: Randomized Controlled Trial of Computerized Cognitive Training in Patients With Atrial Fibrillation With Cognitive Impairment But Without Dementia
Brief Title: Atrial Fibrillation Follow-up Investigation to Recover Memory and learnING Trial
Acronym: AFFIRMING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Wispirit Technology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Chang sheng Ma, Prof., Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-AFFIRMING
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Impairment; Atrial Fibrillation
MeSH Terms: conditions — Cognitive Dysfunction; Atrial Fibrillation | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive training (Experimental)
  Interventions: Behavioral: cognitive training
- active control (Active Comparator)
  Interventions: Behavioral: active control

INTERVENTIONS:
Behavioral: cognitive training — tablet-based cognitive training for 12 weeks, 30 minutes each time, at least 5 times a week
  Arms: cognitive training
Behavioral: active control — tablet-based cognitive training tasks with weak or no difficulty changes, 5 times a week, 30 minutes each time for 12 weeks
  Arms: active control

SUMMARY:
The objective of the study is to evaluate the effectiveness of cognitive training in people with atrial fibrillation and cognitive decline over 12-week cognitive training. Moreover, the investigators will explore whether the training effect can be maintained.

DETAILED DESCRIPTION:
Introduction: Cognitive impairment is a clinical condition characterized of a reduction in memory and/or other cognitive processes that are insufficiently severe to be diagnosed as dementia.The prevalence of dementia among people over 65 years old in China is 5.14% , while the prevalence of mild cognitive impairment is 20.8%. The risk of cognitive impairment and dementia in patients with atrial fibrillation is significantly higher than that those in the same age group, even after adjusted stroke and other common risk factors such as hypertension and diabetes. At present, the effectiveness of cognitive training in patients with atrial fibrillation complicated with cognitive impairment is not clear.

Objectives: The objective of the study is to evaluate whether cognitive training could lead cognitive improvement in patients with cognitive impairment and atrial fibrillation.

Patients and Methods: The proposed study is a double blinded, randomized and controlled trial that will include 200 patients with cognitive impairment and atrial fibrillation. The groups will be randomized to either intervention or active-control group. Both groups will receive computerized cognitive training performed for 30 minutes x 5 times/week over 12 weeks. A neuropsychological assessment will be administered at baseline and week 12 and 24 after the intervention. The structural and functional MRI will be performed at baseline and week 12 after intervention for a sub-study on the effect of cognitive training on brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years;
2. Completion of 6 or more years of education;
3. Atrial fibrillation confirmed by ECG ;
4. Complain of memory decline within 1 year;
5. The score of any cognitive domain in the processing speed, episodic memory, working memory, and visual-spatial tested by the Basic Cognitive Ability Assessment (BCAT) is 1SD less than the average of the normal population;
6. Agree to receive cognitive function testing and randomization, be able to receive follow-up as required

Exclusion Criteria:

1. Unable to complete the test due to vision, hearing and other problems;
2. Dementia or MMSE Scale ≤ 20;
3. Alcohol abuse or taking drugs that affect cognitive function (antihistamines, antipsychotics);
4. Cannot master the method of cognitive training tool after 2 times, 1 hour each time training instruction;
5. Planned atrial fibrillation ablation within 3 months or received ablation in the last 3 months;
6. CHA2DS2-VASc score ≥ 2 (for female ≥ 3), but refuses anticoagulation or has anticoagulation contraindications;
7. General anaesthesia in the last 3 months;
8. A history of stroke and head injury in the last 6 months;
9. Past history of Parkinson's disease, schizophrenia, and epilepsy;
10. Previous neurosurgery or a history of head tumor;
11. Contraindications for MRI examination: such as metal implantation, claustrophobia, etc.;
12. No family members to assist the patients to do the training course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
global cognitive change in 12 weeks | 12 weeks after randomization
  The percentage of patients whose global cognitive function measured at 12 weeks after intervention improves 0.67 SD compared to that measured at baseline by basic cognitive ability test (BCAT)

SECONDARY OUTCOMES:
global cognitive change in 24 weeks | 24 weeks after randomization
  The percentage of patients whose global cognitive function improved at 24 weeks
domain cognitive change | 12 weeks, 24 weeks after randomization
  The percentage of patients whose cognitive function improved in any domain at 12 weeks and at 24 weeks;
cognitive score change | 12 weeks, 24 weeks after randomization
  Changes in global cognitive function scores at 12 weeks and at 24 weeks
self-efficacy scores | 12 weeks, 24 weeks after randomization
  Changes in the patient's self-efficacy scores compared with baseline at 12 weeks and at 24 weeks. The General Self-Efficacy scale ranged from 10 to 40, and higher scores mean better self-efficacy.
quality of life scores | 12 weeks, 24 weeks after randomization
  Changes in the patient's quality of life scores compared with baseline at 12 weeks and at 24 weeks. quality of life will be measured using EQ-5D-3L(EuroQol 5-Dimensional 3 level version).
anxiety and depression scores | 12 weeks, 24 weeks after randomization
  Changes in the patient's anxiety and depression scores compared with baseline at 12 weeks and at 24 weeks. Anxiety status will be measured using the GAD-7 questionnaire which ranges from 0 to 21, with a higher score representing more anxiety. Depression status will be measured using the PHQ-9 questionnaire which ranges from 0 to 27, with a higher score representing more depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Jia J, Zhou A, Wei C, Jia X, Wang F, Li F, Wu X, Mok V, Gauthier S, Tang M, Chu L, Zhou Y, Zhou C, Cui Y, Wang Q, Wang W, Yin P, Hu N, Zuo X, Song H, Qin W, Wu L, Li D, Jia L, Song J, Han Y, Xing Y, Yang P, Li Y, Qiao Y, Tang Y, Lv J, Dong X. The prevalence of mild cognitive impairment and its etiological subtypes in elderly Chinese. Alzheimers Dement. 2014 Jul;10(4):439-447. doi: 10.1016/j.jalz.2013.09.008. Epub 2014 Jan 10. PMID 24418053
- [Background] de Bruijn RF, Heeringa J, Wolters FJ, Franco OH, Stricker BH, Hofman A, Koudstaal PJ, Ikram MA. Association Between Atrial Fibrillation and Dementia in the General Population. JAMA Neurol. 2015 Nov;72(11):1288-94. doi: 10.1001/jamaneurol.2015.2161. PMID 26389654
- [Background] Chen LY, Norby FL, Gottesman RF, Mosley TH, Soliman EZ, Agarwal SK, Loehr LR, Folsom AR, Coresh J, Alonso A. Association of Atrial Fibrillation With Cognitive Decline and Dementia Over 20 Years: The ARIC-NCS (Atherosclerosis Risk in Communities Neurocognitive Study). J Am Heart Assoc. 2018 Mar 7;7(6):e007301. doi: 10.1161/JAHA.117.007301. PMID 29514809
- [Background] Sherman DS, Mauser J, Nuno M, Sherzai D. The Efficacy of Cognitive Intervention in Mild Cognitive Impairment (MCI): a Meta-Analysis of Outcomes on Neuropsychological Measures. Neuropsychol Rev. 2017 Dec;27(4):440-484. doi: 10.1007/s11065-017-9363-3. Epub 2017 Dec 27. PMID 29282641